CLINICAL TRIAL: NCT01733524
Title: Impact of Pet Ownership on Glycemic Control in Youth With Type 1 Diabetes
Brief Title: Pet Ownership and Glucose Control in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Olga Gupta, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R03HD071263-01 (NIH)
Record Dates: First submitted 2012-11-02; First posted 2012-11-27 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: adolescence; self care
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Picture of a fish (Sham Comparator): Participants will receive a picture of a betta fish.
  Interventions: Behavioral: Picture of a fish
- Pet fish (Active Comparator): Participants will receive a betta fish and the supplies to care for the fish for a one year time period.
  Interventions: Behavioral: Pet Fish

INTERVENTIONS:
Behavioral: Pet Fish — Participants will receive a betta fish and the supplies to care for the fish for a one year time period.
  Arms: Pet fish
Behavioral: Picture of a fish — Participants will receive a picture of a betta fish.
  Arms: Picture of a fish

SUMMARY:
The investigators' long-term goal is to discover novel, inexpensive and feasible strategies to improve the management and well-being of youth with T1DM. The specific objective of this proposal is to quantify the impact of responsible pet ownership on the glycemic control and health related quality of life in youth with T1DM.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) affects 151,000 children and adolescents in the United States. Youth with T1DM are at a high risk for multiple psychosocial co-morbidities including poor health related quality of life (HRQoL) which is linked to medication non-compliance and increased risk for diabetes-related complications. Any reduction in the psychosocial adjustment difficulties related to T1DM could improve the medical outcome of children with T1DM.

Current standards for diabetes management reflect the need to maintain glucose control within a normal range. However, numerous reports indicate that normalization of blood glucose levels is seldom attainable in children and adolescents. Family cohesion, positive coping strategies, younger age of onset, social support and adequate self-regulatory behavior are found to favorably influence glycemic control. One may conclude that the presence of a companion animal, capable of enhancing the positive factors named above, would augment the array of tools available for the successful management of chronic illnesses such as T1DM.

There is a lack of studies assessing the impact of pet ownership on the health and well-being of adolescents. The process of caring for, loving and being loved by a companion animal could offer direct and/or indirect benefits to the HRQoL in children with T1DM. To the investigators' knowledge, there are no studies examining the impact of pet ownership on glycemic control and HRQoL in youth with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* 10 to 18 years
* diagnosed with type 1 diabetes for at least 12 months
* poor diabetes control as defined by having a hemoglobin A1c value > 8%

Exclusion Criteria:

* type 2 diabetes
* developmental delay
* current participation in another study that may impact glycemic control

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 12 months
  Hemoglobin A1c values

SECONDARY OUTCOMES:
HRQoL | 9 months
  Generic and diabetes-specific health related quality of life
Self Management of Diabetes in Adolescents | 12 months
  Self management of diabetes in adolescence questionnaire

OTHER OUTCOMES:
Health care burden | 12 months
  Number of visits to the Emergency Department and inpatient hospitalizations for poor glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Olga T Gupta, MD, Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States